CLINICAL TRIAL: NCT06914544
Title: Hypofractionated Radiosurgery for Localised Prostate Cancer (HYPOSTAT-III)
Acronym: HYPOSTAT-III
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: University of Luebeck (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARO-2024-3; DRKS00036292 (Registry Identifier: DRKS - Deutsches Register Klinischer Studien)
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; SBRT; CyberKnife; Radiosurgery; HYPOSTAT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypofractionated Radiosurgery (Experimental): 3 fractions with 9.5-10.5 Gy, total dose 28.5-31.5 Gy
  Interventions: Radiation: Hypofractionated Radiosurgery

INTERVENTIONS:
Radiation: Hypofractionated Radiosurgery — Image-guided stereotactic Linac based RT preferable with "dedicated radiosurgery system" such as CyberKnife

SUMMARY:
Hypofractionated radiosurgery with 5 fractions is considered standard of care for localized prostate cancer. The investigators initiated this multicenter phase II prospective trial to analyse feasibility (toxicity) of hypofractionated radiosurgery with 3 fractions in patients with localised prostate cancer under the hypothesis that the ratio of patients with late GU and GI toxicity ≥ grade 2 after 1 year amounts to 8.4% and 1.3% and is significant lower than 16.4% and 5.7% currently.

DETAILED DESCRIPTION:
Experimental radiosurgery of the prostate with 3 fractions each with 9.5 -10.5 Gy (total application rate of 28.5-31.5 Gy) based on risk grading.

Planned visits are: Baseline, visits at every radiation day and four follow ups (4-6 weeks, 3 months, 6 months and one year after last day of radiation).

ELIGIBILITY:
Inclusion Criteria:

* Localised, histopathologically confirmed Prostate Cancer (cT1-T2c N0 M0)
* Gleason-grade ≤7, ISUP Grade Group 1-3
* Guideline-based staging
* Age ≥ 18 years
* PSA < 20 ng/ml
* Volume of the prostate < 80 cm³
* IPSS-Score ≤ 12
* Written informed consent

Exclusion Criteria:

* History of prior pelvic radiotherapy
* Previous transurethral resection, laser enucleation or prostate ablation
* Contraindication to MRI or Fiducial marker implantation (e.g. gold allergy)
* Relevant comorbidity thought to adversely affect treatment compliance
* Legal incapacity or lack of informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
GU and GI Toxicity | 12-15 months after radiotherapy
  Late toxicity measured with Radiation Therapy Oncology Group-(RTOG)-Score

SECONDARY OUTCOMES:
Acute toxicity | Through study completion
  Acute toxicity analysed by Adverse Event (AE)- and Serious Adverse Event (SAE)-reports
PSA | At the time of inclusion and 1, 3, 6-9 and 12-15 months after radiotherapy
  Prostate Specific Antigen (PSA)
IPSS | Screening and 3, 6-9 and 12-15 months after radiotherapy
  International Prostate Symptom Score (IPSS) on a scale 0-35 with lower being better
Quality of Life Score | At the time of inclusion and 12-15 months after radiotherapy
  EORTC Quality of Life Questionnaire (QLQ) C30 on a scale 0-100 with higher being better
Decision Regret Score | At the time of inclusion and 12-15 months after radiotherapy
  Decision Regret Score on a scale 0-100 with lower being lower regret

CONTACTS AND LOCATIONS:
Overall Officials: David Krug, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (6):
- Germany (6):
  - Saphir Radiosurgery Center Frankfurt am Main, Frankfurt am Main, Hesse
  - University Hospital Frankfurt, Frankfurt am Main, Hesse
  - European Radiosurgery Center Munich, Munich, Hesse
  - Saphir Radiosurgery Center Norther Germany, Kiel, Schleswig-Holstein
  - University Medical Center Schleswig-Holstein, Kiel, Schleswig-Holstein
  - CyberKnife Centrum Mitteldeutschland, Erfurt, Thuringia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Krug D, Imhoff D, Haidenberger A, Hessler N, Schafer J, Huttenlocher S, Chatzikonstantinou G, Furweger C, Ramm U, Konig IR, Chun F, Staehler M, Rodel C, Muacevic A, Vonthein R, Dunst J, Blanck O. Robotic stereotactic body radiotherapy for localized prostate cancer: final analysis of the German HYPOSTAT trial. Strahlenther Onkol. 2023 Jun;199(6):565-573. doi: 10.1007/s00066-023-02044-2. Epub 2023 Feb 9. PMID 36757424